CLINICAL TRIAL: NCT05555056
Title: Enhancing the Effectiveness of Cognitive Behavioral Therapy Using Non-invasive Brain Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Winnipeg Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS25578
Record Dates: First submitted 2022-09-20; First posted 2022-09-26 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Depression; Anxiety; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Thirty participants among those who are enrolled in the parent clinical trial will be recruited. Participants will receive 5-week CBTm treatment and a battery of psychological assessment as part of the parent clinical trial. Individuals enrolled in the current study will receive daily HD-tDCS during the period of CBTm treatment (5-week). Half of the individuals will receive real stimulation and the other half will receive sham stimulation. Participants will be scanned with MRI before and after the 5-week treatment. EEG data will be collected before (10 minutes), during (20 minutes) and after (20 minutes) each HD-tDCS session .
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham stimulation mode will be used in the HD-tES machine. For sham stimulation, the current will be applied for 30 seconds ramp-up followed by 30 seconds ramp-down, and thus no active stimulation will be administered except for the initial and last 1 minutes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Stimulation (Active Comparator): MxN-9 HD-tES Stimulator (Soterix Inc.) will be used to deliver direct current (High-Definition Transcranial Direct Current Stimulation) to the target brain areas via electrodes and conducive gels. A constant current will be applied for 20 minutes with peak current of 2 mA. The 9 electrodes (8 channels + 1 ground) positions and current intensity have been determined based on computer simulation using HDTargets software (Soterix Inc.) that results in maximum focal current on the left VLPFC (x=-50, y=+26, z=+8) and the PCC (x=1, y=-61, z=38) with inward field orientation.
  Interventions: Device: MxN-9 HD-tES Stimulator (Soterix Inc.)
- Inactive Stimulation (Sham Comparator): The current will be applied for 30 seconds ramp-up followed by 30 seconds ramp-down, and thus no active stimulation will be administered except for the initial and last 1 minutes of 20 minute stimulation duration.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: MxN-9 HD-tES Stimulator (Soterix Inc.) — Patients will be stimulated with high definition transcranial direct current stimulation (HD-tDCS) for 5 weeks (every weekdays; one session per day). In each session, a constant current at 2mA will be passed on the target brain areas for 20 minutes.
  Arms: Active Stimulation
Device: Sham Stimulation — The same stimulation protocol will be used as in Active stimulation except that a sham mode will be selected in the stimulator machine.
  Arms: Inactive Stimulation

SUMMARY:
The purpose of the proposed study is to examine if a repeated treatment of High Definition Transcranial Direct Current Stimulation (HD-tDCS) can increase the functional connectivity between the left ventrolateral prefrontal cortex and posterior cingulate, which may further enhance the effects of cognitive behavioral therapy with mindfulness classes.

ELIGIBILITY:
Inclusion Criteria:

* all patients who have agreed to participate in virtual mental health treatment at health care sites throughout Manitoba. Eligible participants will be those enrolled in a range of mental health programs, including CBT, DBT, virtual hospital wards, and group-based treatment (e.g., CBTm, Managing Difficult Emotions, etc). The target population will also include providers and decision makers offering virtual mental health programs. Individuals must meet the following criteria to be eligible to participate in the study: 1) must be a patient/client enrolled in a virtual mental health program OR a provider/decision maker offering a virtual mental health program, and 2) located within Manitoba

Exclusion Criteria:

* contraindication for MRI (e.g., metallic implants and claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Functional Connectivity | Change from Baseline Functional Connectivity after 5 month HD-tDCS/CBTm treatment
  Functional Connectivity between the targeted brain regions measured by resting state fMRI (level of synchronous fMRI signal, standardized)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada